CLINICAL TRIAL: NCT04860492
Title: A Randomized, Double-blind, Placebo-controlled Study of Agropyron Repens, Mannitol and Magnesium Supplement for the Treatment of Calcium Oxalate Upper Urinary Tract Stones: The AMMOS Study
Brief Title: The Impact of Renalof® Dietary Supplement on Upper Urinary Tract Stone Volume
Acronym: AMMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Sountoulidis Petros, Assistant Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Agropyron-1
Record Dates: First submitted 2021-04-13; First posted 2021-04-27 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Calculus of Upper Urinary Tract (Disorder)

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomization sequence will be computer-generated by the study coordinating team
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renalof (Active Comparator): Patients will be given and, advised to take Renalof tablets 325mg three times a day for 90 days
  Interventions: Dietary Supplement: Renalof 325mg
- Placebo (Placebo Comparator): Patients will be given and, advised to take Placebo three times a day for 90 days
  Interventions: Dietary Supplement: Renalof 325mg

INTERVENTIONS:
Dietary Supplement: Renalof 325mg — RENALOF® is a preparation that contains active Agropyron repens extract. It is designed with specific antioxidant compounds triggered by a bio-catalyst process that enables improved control of the production mechanism of anti-stress molecules. RENALOF® contains extracts of couch grass (triticin, potassium salts, agropyron, silicic salt, inositol, vanillin, saponin, mucilage, iron, and others trace elements), mannitol, corn starch and magnesium silicate. The magnesium in RENALOF® inhibits stone formation by inhibition of growth of crystals and aggregation.

SUMMARY:
Following informed consent, all recruited patients will have a baseline non-contrast CT scan performed at the radiology department of "G. Gennimatas" hospital and reported by the same dedicated uroradiologist for evaluation of stone volume, location, and consistency. All patients will also have a free flow mid-stream urinalysis and culture before randomization.

The level of pain related to stones will be evaluated in all patients with the VAS tool completed before commencement of treatment and at the end of the study.

Patients with a DJ stent at study entry will also complete the mini-Ureteral Stent Symptoms Questionnaire (m-USSQ) and the PUF questionnaire completed one week into study, before commencement of treatment and at the end of the study after taking either RENALOF® or placebo. Patients with a DJ stent in situ at study entry, will have both ends of the DJ cut and send for culture during scheduled DJ stent change. Approximately 90 days after recruitment, all patients will have a follow up CT scan, done at "G. Gennimatas" hospital radiology department and evaluated by the same dedicated uroradiologist , and a mid-stream urinalysis and culture. Patients with a DJ in situ will have their catheters changed and cut ends from the distal and proximal stent coils of the removed DJ stents will be send for culture and sensitivity analysis. All patients will complete the VAS and the cohort of patients with DJ stents will complete both the mini-USSQ and PUF questionnaires.

During the study period patients will be instructed to report to the research team any cases of upper or lower urinary tract infection documented with a positive urine culture and any treatment related adverse events.

DETAILED DESCRIPTION:
A total of 82 patients with renal stone or ureteral stones measured on a CT scan performed no later than 1 month prior to randomization, will be recruited in the study. Full medical history as well as demographic data and relevant medical treatment will be recorded in all eligible patients, followed by a detailed physical examination.

All eligible patients who have read and signed the study consent form will be randomized to either RENALOF® or placebo.

The randomization sequence will be computer-generated by the study coordinating team. Randomization will be performed before enrolment of the first patient.

Both the investigators and the study participants will be blinded to the treatment received (RENALOF® or placebo). Following randomization, the participants will be given prefilled non-labelled boxes containing either active drug (RENALOF®) or placebo. The pills in all boxes will be visually identical in size, weight and shape. Each box will have a tag with a unique code. A list of all dispersed coded boxes and the type of drug each box contains (RENALOF® or placebo) will be kept sealed by the study coordinator until the end of the study. Only at the end of the study period the research team will be unblinded to the treatment each patient had received.

The study will be carried out in prespecified time-points, which are listed below:

Point 0 (P0): Screening visit and randomization:

Participants will provide a written informed consent before enrolment. A full medical history will be recorded including medications, interventions for upper tract stones (ESWL, URS, PCNL), medical treatment for stones, history of spontaneous stones passage. Findings on clinical examination and patient demographic characteristics (body weight, height, body mass index (BMI) will be recorded.

The size, number and location of stones on CT scan will be recorded along with any other relevant finding (horseshoe kidney, UPJ obstruction, duplicate collecting system, ureteric stricture etc.). The location, size, surface area and volume of each stone will be calculated and recorded as well as the total stone surface area and stone volume for each patient. All CT studies will be evaluated and stone parameters will be estimated by the same independent dedicated certified radiologist using the Invesalius computer software.

All patients will have a baseline Urea and electrolytes (U and E) blood test, free flow random sample urinalysis and culture. U and E will include serum creatinine, sodium, potassium, calcium and albumin. Parathyroid hormone will also be assessed to confirm or exclude hyperparathyroidism. Urinalysis includes pH, specific weight, sodium, calcium, oxalate, uric acid, citrate and magnesium. Urine culture tests for the possibility of a urinary tract infection (UTI) and if necessary, sensitivity will be carried out which will help treatment.

Patients with indwelling DJ stents will have their stents changed under local anesthesia. In order to reduce patient discomfort and stent related symptoms (SRS) the stent length for each patient will be estimated on the basis of individual patient's height as follows: height < 175 cm will receive a 22F stent, > 175 cm < 190 cm will receive a 24 F stent and patients taller than 190 cm will have a 26F stent. Care will be taken that the loop of the stents in the bladder does not cross the midline. The distal and proximal ends of the stent will be sent for culture. Patients with DJ stents will complete a m-USSQ and a PUF questionnaire 2 weeks following stent insertion or stent change. This will be done in order to avoid bias as patients will have this procedure done under local anesthesia.

Patients will then be randomized and 3 unlabeled boxes containing a total of 120 pills (3-month supply) of either active treatment (RENALOF®) or placebo will be dispersed. The patients will be asked to take 3 pills daily for 90 days.

Point 1 (P1): End of the 90-day RENALOF® treatment All participants will have a follow up CT scan. The location, size, surface area and volume of each stone will be calculated and recorded as well as the total stone surface area and stone volume for each patient. The findings will be compared to those of the baseline CT scan. Estimation of all stone parameters (location, size, surface area, stone volume) will be done by the same radiologist as in the screening visit in order to avoid interobserver variability. Incidences of spontaneous stone passage will be recorded.

All patients will have a repeat free flow urinalysis and culture and complete a VAS.

Patients with DJ stents will have their stents changed and the stent ends will be sent for culture and sensitivity. Patients with stents will complete a m-USSQ and PUF questionnaire. Incidences of UTIs (with a positive urine culture) during the study period will be recorded. Treatment related adverse events and drop-out rates will be recorded.

Once final assessment of all recruited patients has been completed, researchers will be unblinded to the type of treatment each patient has received (RENALOF® or placebo). The patients will then form 2 groups (group A, n = 41, those who received RENALOF®; and group B, n = 41, those who received placebo) and the groups will be compared for primary and secondary study endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Upper urinary tract stones
3. Stone density > 500 HU on CT (Mean Hounsfield Units of the largest stone)
4. Ability to understand and provide a written informed consent to participate in the study

Exclusion Criteria:

1. Staghorn stones occupying renal calyces and pelvis
2. Stone composition other than calcium, indirectly assessed or determined using the Hounsfield stone density units (a Mean Hounsfield score of < 500 units will be considered)
3. Use of other urinary urinary stone treatments
4. Use of magnesium supplementation
5. Chronic kidney disease (CKD) with eGFR<30 ml/sec
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Stone volume | 90 days
  Stone volume (measured in mls) will be calculated using a dedicated software

SECONDARY OUTCOMES:
Stent-related symptoms score in the cohort of patients with DJ stents. | 90 days
  Symptoms score will be assessed using the mini-Ureteral Stent Symptoms Score (m-USSS). The Mini Ureteral Stent Symptoms Questionnaire (mini-USSQ) is a validated, simplified, and shorter version of the 38 item Ureteral Stent Symptoms Questionnaire. It has 8 questions and a maximum of 77 points for women and 87 for men with maximum values showing worst symptoms.
Overactive Bladder (OAB) Symptoms score | 90 days
  OAB scores will be assessed by the Pelvic Pain and Urgency-Frequency (PUF) questionnaire.The Pelvic Pain and Urgency/Frequency Patient Symptoms Scale (PUF) is an 8 question instrument used to assess pelvic symptoms. Scores range from 0 to 35 points with 35 being the worst feeling of pelvic related discomfort.
Pain level | 90 days
  Pain scores will be assessed by the Visual Analogue Score (VAS).The Visual analogue score (VAS) is an tool which is used to determine pain on a level from 1 to 10 shown diagrammatically. No pain is 1 on the VAS score and excessive pain is indicated with a 10 on the scale.
Microbial growth of double J stents in the cohort of patients with DJ stents. | 90 days
  the proximal and distal ends of the removed double J stents will be sent for culture
Incidence of documented urinary tract infections | 90 days
  patients will be asked to report any urinary tract infections (defined as symptoms of a UTI and a positive urine culture)

CONTACTS AND LOCATIONS:
Overall Officials: Petros Sountoulides, M.D, Phd, Principal Investigator — Aristotle Univeristy
Locations (1):
- G. Gennimatas Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No